CLINICAL TRIAL: NCT07228910
Title: Relationship Between Dysfunctional Breathing, Respiratory Patterns, and Performance Anxiety in Music Students
Brief Title: Respiratory and Anxiety Status of Music Students
Status: Not yet recruiting | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Erhan KIZMAZ, Assistant professor, Pamukkale University
Other Study IDs: Music
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Dysfunctional Breathing; Breathing Patterns
Keywords: Dysfunctional breathing; Breathing patterns; Music students; Music performance anxiety

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to determine the prevalence and patterns of dysfunctional breathing (DB) among music students and to investigate its relationship with music performance anxiety (MPA). Dysfunctional breathing, also known as a breathing pattern disorder, refers to maladaptive respiratory patterns not explained by medical conditions such as asthma and is associated with symptoms like hyperventilation, poor breathing control, and abnormal respiratory mechanics. Given that MPA is common among musicians and often accompanied by symptoms such as palpitations, tremor, and shortness of breath, this study explores whether DB contributes to or is influenced by performance-related anxiety in this population.

DETAILED DESCRIPTION:
Dysfunctional breathing (DB) represents a spectrum of maladaptive respiratory patterns that cannot be explained by an underlying medical condition. It may involve biomechanical, biochemical, or psychophysiological components, including abnormal breathing mechanics, altered carbon dioxide regulation, and stress-related breathing irregularities. Previous research has suggested that DB can exacerbate symptoms in conditions such as asthma, migraine, orofacial pain, and temporomandibular disorders.

Music performance anxiety (MPA), a common issue among music students and professional musicians, manifests through both psychological and physiological symptoms. Among these, respiratory complaints such as dyspnea, breath-holding, or hyperventilation are frequently reported. Despite this, the potential overlap between DB and MPA has not been adequately investigated.

This cross-sectional study will assess 233 music students using validated self-report questionnaires to evaluate dysfunctional breathing patterns and levels of music performance anxiety. The study seeks to identify the prevalence of DB in this population and to explore possible associations between breathing dysfunction and anxiety related to musical performance. Findings may contribute to a better understanding of respiratory-related mechanisms underlying performance anxiety and inform preventive or therapeutic strategies for musicians.

ELIGIBILITY:
Inclusion Criteria:

* Being a student of music department
* Playing an instrument for at least 1 year
* Volunteer

Exclusion Criteria:

* Having any respiratory disease (Asthma , COPD etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Music department students from three different universities (Munzur University, Gaziantep University and, Mehmet Akif Ersoy University) will be invited to our study.
Sampling Method: Probability Sample
Enrollment: 233 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Dysfunctional breathing | 15 minutes drom enrollment
  An umbrella term used to describe a harmful adaptation in breathing that cannot be explained by a medical diagnosis such as asthma. The Self Evaluation of Breathing Questionnaire (SEBQ) will be used to assess dysfunctional breathing. The SEBQ is a scale developed to identify the nature of unexplained symptoms commonly reported by individuals with dysfunctional breathing. It was designed to capture all domains of respiratory symptoms, regardless of whether the individual has hyperventilation syndrome. The questionnaire consists of 25 items rated on a 4-point Likert scale ranging from 0 to 3 (0 = never / not true at all, 1 = occasionally / somewhat true, 2 = often / mostly true, 3 = very often / very true). Higher scores indicate a greater degree of breathing dysfunction
Breathing pattern | 15-30 minutes from enrollment
  The Breathing Pattern Assessment Tool (BPAT) will be used to assess breathing pattern. The BPAT is a clinician-administered assessment developed to evaluate breathing pattern disorders. Its validity has been confirmed for screening breathing pattern dysfunction in patients with asthma or unexplained dyspnea. During the assessment, the participant is seated in a chair with back support while the clinician evaluates seven components of the breathing pattern: abdominal and chest wall movements, inspiratory and expiratory sounds, sighing or other signs of air hunger, nasal and oral breathing, breathing rate, and rhythmicity of the pattern. Each item is scored from 0 to 2, yielding a total score ranging from 0 to 14. Higher scores indicate a greater likelihood of breathing pattern disorder. A total score of ≥4 is considered a positive screen, with a sensitivity of 92% and specificity of 75%.
Music performance anxiety | 30-45 minutes from enrollment
  The Kenny Music Performance Anxiety Inventory (K-MPAI) will be used to assess the level and underlying causes of music performance anxiety. T. The inventory consists of 25 items grouped under five subscales: (1) Negative Performance Perception (items 5, 6, 10, 11, 13, 14, 15, 16, 18, 19, 22, 23, 24, 25), (2) Psychological Vulnerability (items 1, 2, 3, 7, 8, 9, 12, 21), (3) Somatic Anxiety (item 4), (4) Personal Control (item 17), and (5) Physiological Vulnerability (item 20). Each item is rated on a 7-point Likert scale ranging from 0 (strongly disagree) to 6 (strongly agree), yielding a total score between 0 and 150. Scores of 105 and above indicate high music performance anxiety, whereas scores of 45 and below indicate low anxiety levels.

CONTACTS AND LOCATIONS:
Overall Officials: Erhan KIZMAZ, PhD, Principal Investigator — University of Gaziantep

IPD SHARING:
Plan to Share IPD: Undecided